CLINICAL TRIAL: NCT05908591
Title: SLEEP: Sleep Disordered Breathing, Endothelial Function, and Adverse Events in Pregnancy
Brief Title: Sleep Disordered Breathing, Endothelial Function, and Adverse Events in Pregnancy
Acronym: SLEEP
Status: Recruiting | Type: Observational
Sponsor: University of Alberta (Other)
Responsible Party: Sponsor
Other Study IDs: Pro00110658
Record Dates: First submitted 2023-05-17; First posted 2023-06-18 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Pregnancy Related; Sleep-Disordered Breathing
Keywords: Cardiovascular Health
MeSH Terms: conditions — Sleep Apnea Syndromes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This is a prospective longitudinal cohort study whereby pregnant individuals are asked to complete an 8-day testing protocol to measure their sleep and cardiovascular health at two timepoints during pregnancy.

DETAILED DESCRIPTION:
The goal of this observational study is to examine the effect of sleep disordered breathing on the health of the heart and blood vessels of the mother during pregnancy. The main questions it aims to answer are:

* Is sleep disordered breathing associated with impaired the function of the heart and blood vessels in pregnancy?
* Is higher levels of physical activity associated with a reduced risk of sleep disordered breathing in pregnancy?

Participants will complete an 8 day long study protocol at two time points during pregnancy (20-24 weeks gestation and 28-36 weeks gestation). During each testing period they will be asked to:

* Complete one night of at-home sleep testing and and one night of overnight vital signs monitoring (ambulatory blood pressure and heart rate monitoring devices)
* Wear two accelerometers and complete a 7-day sleep log
* Complete a set of questionnaires
* Visit the laboratory for a fasted blood draw and ultrasound assessment of their cardiovascular health (resting heart rate and blood pressure, flow mediated dilation and pulse wave velocity tests)

Participants will also be asked to complete a short follow-up survey in the postpartum period.

ELIGIBILITY:
Inclusion Criteria:

* over 18 years of age
* pregnant (20-24 weeks gestation at enrollment)

Exclusion Criteria:

* worked shift work past 11pm in the previous month
* previously diagnosed with a sleep disorder by a physician

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Pregnant individuals with and without symptoms of sleep disordered breathing.
Sampling Method: Non-Probability Sample
Enrollment: 109 (Estimated)
Dates: Start 2023-01-01 (Actual); Primary Completion 2027-04-18 (Estimated); Study Completion 2027-04-18 (Estimated)

PRIMARY OUTCOMES:
Endothelial Function | 20-24 weeks and 28-36 weeks gestation
  The investigators will assess endothelial function using flow mediated dilation

SECONDARY OUTCOMES:
Cardiovascular Function - arterial stiffness with pulse wave velocity | 20-24 weeks and 28-36 weeks gestation
  The investigators will measure arterial stiffness using pulse wave velocity of the carotid and femoral arteries
Cardiovascular Function - arterial stiffness with beat-by-beat blood pressure | 20-24 weeks and 28-36 weeks gestation
  The investigators will measure arterial stiffness using beat-by-beat blood pressure from the finger.
Cardiovascular Function - ambulatory blood pressure | 20-24 weeks and 28-36 weeks gestation
  Blood pressure will be collected every 30 minutes during a 24-hour period using an ambulatory blood pressure monitor.
Cardiovascular Function - resting blood pressure | 20-24 weeks and 28-36 weeks gestation
  Beat-by-beat blood pressure will be collected at rest.
Cardiovascular Function - heart rate | 20-24 weeks and 28-36 weeks gestation
  Heart rate will be assessed by 3-lead ECG collected during sleep and at rest.
Cardiovascular Function - arrythmias | 20-24 weeks and 28-36 weeks gestation
  Presence of arrythmias will be assessed by 3-lead ECG collected during sleep and at rest.
Maternal outcome - dietary intake | 20-24 weeks and 28-36 weeks gestation
  Participants will complete two 3-day food logs.
Fasted blood sample - blood viscosity | 20-24 weeks and 28-36 weeks gestation
  Fasted blood samples will be analyzed using a viscometer.
Fasted blood sample - presence of inflammatory markers | 20-24 weeks and 28-36 weeks gestation
  Fasted blood samples will be analyzed for C-reactive protein.
Fasted blood sample - sex hormone levels | 20-24 weeks and 28-36 weeks gestation
  Fasted blood samples will be analyzed for sex hormone levels (estrogen, progesterone, testosterone).
Fasted blood sample - metabolic | 20-24 weeks and 28-36 weeks gestation
  Fasted blood samples will be analyzed for glucose and insulin concentration.
Maternal outcomes - delivery | 2 months postpartum
  Participants will provide the investigators with information regarding delivery and pregnancy complications (gestational diabetes, pregnancy induced hypertension, preeclampsia).
Fetal outcomes at delivery - infant sex | 2 months postpartum
  Participants will provide the investigators with information regarding infant sex.
Fetal outcomes at delivery - birth weight | 2 months postpartum
  Participants will provide the investigators with information regarding infant birth weight.
Fetal outcomes at delivery - birth length | 2 months postpartum
  Participants will provide the investigators with information regarding birth length.
Fetal outcomes at delivery - gestational age | 2 months postpartum
  Participants will provide the investigators with information regarding gestational age at delivery.
Fetal outcomes at delivery - birth mode | 2 months postpartum
  Participants will provide the investigators with information regarding birth mode.
Fetal outcomes at delivery - apgar score | 2 months postpartum
  Participants will provide the investigators with information regarding infant apgar score at delivery.
Fetal outcomes at delivery - time spent in NICU | 2 months postpartum
  Participants will provide the investigators with information regarding infant time spent in neonatal intensive care unit (NICU).
Maternal outcome - amount of activity | 20-24 weeks and 28-36 weeks
  Participants will wear two accelerometers to measure the amount of physical activity performed.
Maternal outcome - Mood - State-Trait Anxiety Inventory | 20-24 weeks and 28-36 weeks
  Participants will complete the State-Trait Anxiety Inventory to measure mood.
Maternal outcome - Mood - Edinburgh Postnatal Depression Scale | 20-24 weeks and 28-36 weeks
  Participants will complete the Edinburgh Postnatal Depression Scale to measure mood.

CONTACTS AND LOCATIONS:
Locations (1):
- Program for Pregnancy and Postpartum Health, University of Alberta, Edmonton, Alberta, Canada